CLINICAL TRIAL: NCT00932165
Title: Special Investigation For Patients With Renal And/Or Hepatic Disorders On Aromasin (Regulatory Post Marketing Commitment Plan)
Brief Title: Special Investigation For Patients With Renal And/Or Hepatic Disorders On Aromasin
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A5991078
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Results first posted 2010-06-24 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exemestane: Patients taking Exemestane Tablets.
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Exemestane — Aromasin® Tablets 25mg, depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. " The usual adult dose is 25 mg of exemestane administered orally once daily after a meal."
  Other Names: Aromasin

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Exemestane (Aromasin) should be registered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with postmenopausal breast cancer (including ovariectomy etc.).

Exclusion Criteria:

* Patients cannot be evaluated.For example, not administered Exemestane (Aromasin).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A5991078 prescribes the Exemestane (Aromasin).
Sampling Method: Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2004-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991078&StudyName=Special%20Investigation%20For%20Patients%20With%20Renal%20And/Or%20Hepatic%20Disorders%20On%20Aromasin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients need to be administered Exemestane (Aromasin) in order to be enrolled in the surveillance.
Groups:
- Exemestane: Exemestane(Aromasin) as prescribed by subject's physician
Period: Overall Study
Arm/Group | Exemestane
Started | 451
Completed | 450
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exemestane
Number analyzed (Participants) | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 269
  >=65 years | 181
Age Continuous [Mean (Standard Deviation); unit: years] | 62.67 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 450
  Male | 0
Region of Enrollment [Number; unit: participants]
  Japan | 450

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Unexpected Adverse Drug Reaction
Description: Adverse drug reaction that is not included in the "precautions for use"or "undesirable effects" section in the package insert (same as Local Product Document).
Time Frame: 24 weeks
Population: Safety analysis population included all enrolled subjects who had received at least 1 confirmed, administration of exemestane.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 450
participants
  Gastritis | 2
  Hyperlipidaemia | 1
  Angina pectoris | 1
  Asthenia | 1
  Dyspepsia | 1
  Abdominal discomfort | 1
  Constipation | 1
  Hiatus hernia | 1
  Erythema | 1
  Urticaria | 1

2. Primary Outcome: Number of Participants With Factors Considered to Affect the Safety and/or Efficacy of Exemestane
Description: Assessment of factors likely to affect the safety and/or efficacy: reason for Exemestane use (primary progressive breast cancer, relapsed breast cancer or postoperative adjuvant therapy)and past history (presence or absence of at least one disease).
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Exemestane: All the patients whom an investigator prescribes the first Exemestane(Aromasin) should be registered.
Arm/Group | Exemestane
Number analyzed (Participants) | 450
participants
  Primary Progressive Breast Cancer | 126
  Post-operative Adjuvant Therapy | 324
  Past history (nothing at all) | 372
  Past history (presence of at least one disease) | 68
  Unknown history | 10

3. Secondary Outcome: Number of Participants With Adverse Drug Reaction for Subjects With Hepatic Dysfunction
Description: The participants who were diagnosed by the investigator as the participants with hepatic dysfunction, and observed for safety information.
Time Frame: 24 weeks
Population: Subjects with hepatic Dysfunction.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 54
participants
  Hot flush | 1
  Abdominal discomfort | 1
  Rash | 1
  Arthralgia | 1
  Musculoskeletal stiffness | 1
  Aspartate aminotransferase increased | 1
  Gamma-glutamyltransferase increased | 1

4. Primary Outcome: Number of Participants With Performance Status Score Based on Eastern Cooperative Oncology Group (ECOG) Factors Considered to Affect the Safety and/or Efficacy of Exemestane
Description: Scale 0; Asymptomatic (Fully active, able to carry on all predisease activities without restriction), 1; Symptomatic but completely ambulatory (Restricted in physically strenuous activity ,ambulatory and able to carry out light or sedentary work), 2 ; Symptomatic, <50% in bed during the day (Ambulatory,capable of all self care, unable to carry out any work activities., 3; Symptomatic, >50% in bed, not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more waking hours), 4; Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair)
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 450
participants
  Asymptomatic | 385
  Symptomatic, completely ambulatory | 47
  Symptomatic, <50% in bed during the day | 9
  Symptomatic, >50% in bed | 6
  Bedbound | 3

5. Primary Outcome: Number of Participants With Adverse Drug Reaction
Description: Confirmation of the number of subjects with treatment related adverse events. All adverse events regardless of causal relationship with Aromasin Tablet at the end of observation period was reported.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 450
participants | 58

6. Secondary Outcome: Number of Participants With Adverse Drug Reaction for Subjects With Renal Dysfunction
Description: The participants who were diagnosed by the investigator as the participants with renal dysfunction, and observed for safety information.
Time Frame: 24 weeks
Population: Subjects with renal Dysfunction.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 50
participants
  Hot flush | 1
  Hepatic function abnormal | 1
  Osteoporosis | 2
  Back pain | 1
  Gamma-glutamyltransferase abnormal | 1

7. Primary Outcome: Number of Tumor Responders in Progressive Breast Cancer or Recurrent Breast Cancer to Exemestane Treatment
Description: Anti-tumor effect was evaluated according to the rules for 'General Rules for Clinical and Pathological Recording of Breast Cancer' (the 15th edition)/Response Evaluation Criteria in Solid Tumors (RECIST) Guideline. Judged as Completed response (CR) or partial response (PR), stable disease (SD) or progressive disease (PD) after the treatment start.
Time Frame: 24 weeks
Population: N = number of participants with tumor response
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 50
participants
  Completed response (CR) | 1
  Partial response (PR) | 5
  Stable disease (SD) | 12
  Progressive disease (PD) | 32

8. Primary Outcome: Number of Post-operative Adjuvant Therapy Participants With Breast Cancer Recurrence Status
Time Frame: 24 weeks
Population: The participants who were evaluated for efficacy of Aromasin for the post-operative adjuvant therapy.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 320
participants
  Recurrence present | 3
  Recurrence absent | 317

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Exemestane
Serious Adverse Events (participants affected / at risk) | 2/450
Other Adverse Events (participants affected / at risk) | 58/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=450)
Angina pectoris (Cardiac disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=450)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hot flush (Vascular disorders) | 4
Gastritis (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 9
Liver disorder (Hepatobiliary disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Asthenia (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 4
Gamma-glutamyltransferase abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.